CLINICAL TRIAL: NCT03913845
Title: The Impact of Retropubic Lidocaine vs Saline on Postoperative Urinary Retention Following Midurethral Sling: A Randomized Placebo Controlled Trial
Brief Title: The Impact of Retropubic Lidocaine vs Saline on Postoperative Urinary Retention Following Midurethral Sling
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West Penn Allegheny Health System (Other)
Collaborators: AHN Research Institute (Unknown)
Responsible Party: Principal Investigator, Lindsay Turner, MD Female Pelvic Medicine, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Retropubic Lidocaine vs Saline
Record Dates: First submitted 2019-03-20; First posted 2019-04-12 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Lidocaine; Epinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 0.5% lidocaine with epinephrine (Experimental): On the day of surgery, the operating room pharmacist will prepare 20 cc of either study drug (0.5% lidocaine with epinephrine 1:200,000) or normal saline with epinephrine 1:200,000) in identical appearing 20cc syringes to be injected retropubically. Our group's routine clinical practice is to inject 20cc of 0.5% lidocaine with epinephrine 1:200,000 retropubically along the path of the midurethral sling trocars. Suburethral injection of local anesthestic will be performed at surgeon discretion. Surgical teams, anesthesia teams and patients will be blinded to allocation assignment. The investigational drug pharmacist will maintain the randomization sequence.
  Interventions: Drug: lidocaine with epinephrine
- Normal saline with epinephrine (Active Comparator): On the day of surgery, the operating room pharmacist will prepare 20 cc of either study drug (0.5% lidocaine with epinephrine 1:200,000) or normal saline with epinephrine 1:200,000) in identical appearing 20cc syringes to be injected retropubically. Our group's routine clinical practice is to inject 20cc of 0.5% lidocaine with epinephrine 1:200,000 retropubically along the path of the midurethral sling trocars. Suburethral injection of local anesthestic will be performed at surgeon discretion. Surgical teams, anesthesia teams and patients will be blinded to allocation assignment. The investigational drug pharmacist will maintain the randomization sequence.
  Interventions: Drug: Normal saline with epinephrine

INTERVENTIONS:
Drug: lidocaine with epinephrine — One of the most commonly used local anesthetic agents in surgical practice is lidocaine. Lidocaine as a local anesthetic is characterized by a rapid onset of action (typically within 2-5 minutes of injection) and intermediate duration of efficacy and thus is often favored in the outpatient setting for pre-incisional injections. Of note, however, its effects general only last up to 2 hours. Epinephrine (adrenaline) vasoconstricts arteries, delaying the resorption of lidocaine, and thus almost doubles the duration of anesthesia.
  Arms: 0.5% lidocaine with epinephrine
Drug: Normal saline with epinephrine — Several mechanisms could explain the inability to void postoperatively, including nerve conduction impairment from anesthesia. Multiple studies have investigated the use of various types of anesthesia and downstream effects on postoperative urinary retention. It is postulated that denervating the regional pelvic nerves for pain control may lead to denervation of the bladder for a transient period of time, block both the afferent and efferent pathways of the voiding mechanism, affect the urethral retro-resistance pressure and impact urethral length thereby contributing to voiding dysfunction postoperatively. The use of normal saline in this setting may have a reduction in rates and duration of postoperative urinary retention following retropubic midurethral sling placement.
  Arms: Normal saline with epinephrine

SUMMARY:
Stress urinary incontinence affects millions of women worldwide and has a profound impact on the quality of life of older individuals, their subjective health status, levels of depression and need for care. Midurethral sling placement was introduced in 1995 and remains the current gold standard for surgical management of SUI. Although the advantages of midurethral sling surgery include its high success and minimally invasive approach, approximately 10-50% of women experience acute postoperative urinary retention and are subsequently sent home with an indwelling foley catheter or clean intermittent self catheterization. Urinary retention is anxiety provoking for most patients and adds morbidity, cost, and increased utilization of healthcare resources. Additionally, catheterization of the urinary tract results in increased risk of urinary tract infection and potential need for antibiotics.

Several recent studies have reported varying rates of postoperative voiding trial success depending on the type of local anesthetic used for hydrodissection; however the data is sparse and invites a more thorough investigation. Furthermore, to the investigators knowledge, no studies have systematically explored dosage or type of agent used intraoperatively on postoperative voiding function. Based on the preliminary data, the investigators hypothesize that patients receiving normal saline compared to a local anesthetic (e.g., lidocaine) will have a reduction in duration of postoperative urinary retention following retropubic midurethral sling placement.

DETAILED DESCRIPTION:
Aim 1: to compare the incidence of urinary retention following retropubic midurethral sling placement in those women receiving normal saline vs lidocaine for retropubic hydrodissection. The investigators will compare rates of failed retrograde voiding trials between patients receiving normal saline to those receiving the same quantity of lidocaine. This will be completed using a standardized retrograde voiding trial 1-2 hours postoperatively (as outlined in "Data and Statistical Methods" below). The investigators hypothesize that patients receiving normal saline compared to a local anesthetic will have a reduction in postoperative urinary retention following retropubic midurethral sling placement.

Aim 2: to assess postoperative pain in women receiving retropubic normal saline vs lidocaine during midurethral sling placement. Postoperatively, subjects will be asked to mark their pain on a VAS scale administered 2 hours and 6 hours following surgery. The initial assessment will be performed by nursing personnel at the time of routine vital sign assessment; the subsequent assessments will be completed by patients with an at-home form through postoperative day #7. Narcotic use will be queried through the electronic medical record as well as with a pain diary administered at time of discharge until postoperative day #7.

Aim 3: to examine differences in patient satisfaction and quality of life following retropubic midurethral sling placement between women receiving retropubic normal saline vs lidocaine at time of midurethral sling placement. Differences in patient satisfaction will be compared using a Likert Scale. Patients will be asked to rate their satisfaction with surgery on a Likert scale (with 1 being the least satisfied and 5 being the most) at their 6 week postoperative follow up visit. The investigators hypothesize that women receiving normal saline for hydrodissection will have improved patient satisfaction as evidenced by higher Likert scores compared to those receiving lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* English speaking
* Competent to give consent

Exclusion Criteria:

* A known intolerance or allergic reaction to local anesthetics
* Planned spinal anesthesia for the procedure
* Planned concomitant prolapse repair other than anterior repair
* Preoperative voiding dysfunction as evidenced by a postvoid residual (PVR) of 150 mL or greater.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
The incidence of urinary retention | This will be completed using a standardized retrograde voiding trial 1-2 hours postoperatively.
  To compare the incidence of urinary retention following retropubic midurethral sling placement in those women receiving normal saline vs lidocaine for retropubic hydrodissection.

SECONDARY OUTCOMES:
Postoperative pain: VAS scale | Subjects will be asked to mark their pain on a VAS scale administered 2 hours and 6 hours following surgery. The subsequent assessments will be completed by patients with an at-home form through postoperative day #7.
  To assess postoperative pain in women receiving retropubic normal saline vs lidocaine during midurethral sling placement. Visual Analog Scale (VAS) pain scales are unidimensional measures of pain intensity that are easily completed and scored. Subjects place an "X" on a 10 centimeter (cm) VAS line at the point that represents their pain intensity. The score is calculated by measuring the distance in millimeters (mm) along the 10 cm line where 0 represents "no pain" and 10 represents "worst pain." Scores range from 0-100mm. They have been widely used in diverse populations to assess pain. VAS pain scores will be used as the outcome measure in this study because they are easy to complete and because they are easily compared to prior studies. The 2 hour VAS score will be completed prior to discharge. The 6 hour VAS score will be returned via mail since patients are routine discharged a few hours after sling surgery.

OTHER OUTCOMES:
Patient satisfaction following surgery: Likert Scale | 6 weeks postoperatively
  To examine differences in patient satisfaction with surgery between women receiving retropubic normal saline vs lidocaine at time of midurethral sling placement. The Likert Scale is the most widely used approach to scaling responses in survey research and contains five tiered responses which users quantify on a visual analogue scale. The administration of such is easily comprehended, provides an effective and clinically relevant means of assessing patient satisfaction, and can readily be used in clinical practice. To determine satisfaction, patients will be asked to rate their satisfaction with surgery on a Likert scale (with 1 being the least satisfied and 5 being the most) at their 6 week postoperative follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Turner, MD, Principal Investigator — Department of Obstetrics and Gynecology, Allegheny Health Network
Locations (4):
- United States (4):
  - AHN Bethel Park Health + Wellness Pavilion, Bethel Park, Pennsylvania
  - AHN Jefferson Hospital, Jefferson Hills, Pennsylvania
  - AHN West Penn Hospital, Pittsburgh, Pennsylvania
  - AHN Wexford Health + Wellness Pavilion, Wexford, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ICOPE guidelines - World Health Organization. https://www.who.int/ageing/publications/guidelines-icope/en/
- [Background] Duenas-Garcia OF, Patterson D, De la Luz Nieto M, Leung K, Flynn MK. Voiding Function After Midurethral Slings With and Without Local Anesthetic: Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2017 Jan/Feb;23(1):56-60. doi: 10.1097/SPV.0000000000000343. PMID 27682748
- [Background] Bracken JN, Huffaker RK, Yandell PM, Handcock T, Higgins EW, Kuehl TJ, Shull BL. A randomized comparison of bupivacaine versus saline during placement of tension-free vaginal tape. Female Pelvic Med Reconstr Surg. 2012 Mar-Apr;18(2):93-6. doi: 10.1097/SPV.0b013e3182436655. PMID 22453319
- [Background] Nilsson CG, Kuuva N, Falconer C, Rezapour M, Ulmsten U. Long-term results of the tension-free vaginal tape (TVT) procedure for surgical treatment of female stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12 Suppl 2:S5-8. doi: 10.1007/s001920170003. PMID 11450979
- [Background] Nilsson CG, Falconer C, Rezapour M. Seven-year follow-up of the tension-free vaginal tape procedure for treatment of urinary incontinence. Obstet Gynecol. 2004 Dec;104(6):1259-62. doi: 10.1097/01.AOG.0000146639.62563.e5. PMID 15572486
- [Background] Mazloomdoost D, Pauls RN, Hennen EN, Yeung JY, Smith BC, Kleeman SD, Crisp CC. Liposomal bupivacaine decreases pain following retropubic sling placement: a randomized placebo-controlled trial. Am J Obstet Gynecol. 2017 Nov;217(5):598.e1-598.e11. doi: 10.1016/j.ajog.2017.07.001. Epub 2017 Jul 8. PMID 28694151
- [Background] Nicolle LE. Catheter associated urinary tract infections. Antimicrob Resist Infect Control. 2014 Jul 25;3:23. doi: 10.1186/2047-2994-3-23. eCollection 2014. PMID 25075308
- [Background] Balakrishnan K, Ebenezer V, Dakir A, Kumar S, Prakash D. Bupivacaine versus lignocaine as the choice of locall anesthetic agent for impacted third molar surgery a review. J Pharm Bioallied Sci. 2015 Apr;7(Suppl 1):S230-3. doi: 10.4103/0975-7406.155921. PMID 26015720
- [Background] Petros PE, Ulmsten UI. An integral theory of female urinary incontinence. Experimental and clinical considerations. Acta Obstet Gynecol Scand Suppl. 1990;153:7-31. doi: 10.1111/j.1600-0412.1990.tb08027.x. PMID 2093278
- [Background] Duckett JR, Patil A, Papanikolaou NS. Predicting early voiding dysfunction after tension-free vaginal tape. J Obstet Gynaecol. 2008 Jan;28(1):89-92. doi: 10.1080/01443610701811837. PMID 18259908
- [Background] Choi S, Mahon P, Awad IT. Neuraxial anesthesia and bladder dysfunction in the perioperative period: a systematic review. Can J Anaesth. 2012 Jul;59(7):681-703. doi: 10.1007/s12630-012-9717-5. Epub 2012 Apr 26. PMID 22535232

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT03913845/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT03913845/ICF_001.pdf